CLINICAL TRIAL: NCT06977542
Title: A Single-Arm, Phase II Clinical Study of Neoadjuvant Therapy With Ivonescimab Combined With Chemotherapy in Patients With Early or Locally Advanced Triple-Negative Breast Cancer
Brief Title: Neoadjuvant Therapy With Ivonescimab Combined With Chemotherapy for Triple-Negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, MD, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-201
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: TNBC, Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Ivonescimab Plus Chemotherapy
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — a PD-1/ VEGF Bispecific Antibody, 20mg/kg, every 2 weeks;
  Chemotherapy : paclitaxel and carboplatin, followed by epirubicin-cyclophosphamide
  Other Names: AK112

SUMMARY:
This study is a multicenter, single-arm, investigator-initiated Phase II clinical trial. Eligible patients with treatment-naive early or locally advanced triple-negative breast cancer (TNBC), clinically staged as Stage II-III, will receive neoadjuvant therapy with ivonescimab in combination with chemotherapy prior to surgery. During the neoadjuvant phase, ivonescimab will be administered for a total of 12 doses. Patients who complete the neoadjuvant treatment and are deemed surgically eligible must undergo definitive surgical intervention.

Following surgery and pathological evaluation by the local pathology department at each participating center, patients will continue to receive adjuvant therapy with ivonescimab for an additional 14 doses, in addition to any subsequent treatment recommended by the investigator according to standard clinical practice.

The primary endpoint of this study is the pathological complete response rate (pCR). Participants will also be followed for secondary endpoints including event-free survival (EFS), disease-free survival (DFS), and distant disease-free survival (DDFS), with a minimum follow-up duration of 2 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 75 years old, female.

  2. Patients with histologically confirmed unilateral primary invasive breast cancer who meet the criteria of clinical stage II （T1cN1M0/T2N0-1M0/T3N0M0）or stage III (T1cN2-N3M0/T2N2-3M0/T3N1-3M0）.

  3. Patients with Triple Negative breast cancer.

  4. According to the RECIST 1.1 criteria, there is at least one measurable objective lesion.

  5. Eastern Cooperative Oncology Group (ECOG) performance score 0-1.

  6. Appropriate haematological, hepatic and renal function : 1) Absolute number of neutrophils (ANC) ≥ 1.5 x 10^9/L; 2) Platelets ≥ 100 x 10^9/L; 3) Hemoglobin ≥ 90 g/L ; 4) White blood cell (WBC) ≥ 3.0×10^9/L and ≤15×10^9/L; 5) Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); 6) AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN; 7) serum creatinine (Cr) ≤1.5×ULN, and creatinine clearance (CrCL) ≥50 mL/min (Cockcroft-Gault equation); 8) Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5 ULN with international normalized ratio (INR) ≤1.5 ULN (not receiving anticoagulation); 9) Serum albumin ≥ 28g/L.10)Left ventricular ejection fraction (LVEF) ≥ 50%.11)Urine test: urinary protein < 2+; If urinary protein ≥ 2+, 24-hour urinary protein quantification must show protein ≤1g.

  7. Subject is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

  8. With good compliance with the planned treatment, are able to understand the follow-up procedures of this study and sigh the informed consent form.

Exclusion Criteria:

* 1. Cancer-related history and treatment history: a. Bilateral breast cancer. b. History of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS). c. History of invasive or metastatic breast cancer. d. Prior surgical resection or biopsy of the primary breast tumor or axillary metastatic lymph nodes before informed consent was obtained.e. Diagnosis of any malignancy within 5 years prior to signing informed consent, except for cured cervical in situ carcinoma, basal cell carcinoma, or squamous cell carcinoma of the skin.f. Systemic chemotherapy, targeted therapy, or local radiotherapy within 1 year prior to signing informed consent. g. Prior treatment with PD-1/PD-L1 antibodies, CTLA-4 antibodies, or other anti-PD-1/PD-L1 immunotherapies. h. Prior systemic treatment with anthracyclines, taxanes, or platinum-based agents for any malignancy.

  2. Concomitant Diseases/History or Treatments: a.Immunodeficiency disease, b. Active or history of autoimmune disease requiring ongoing treatment, c. Known or suspected interstitial pneumonia; d. Severe cardiovascular or cerebrovascular diseases, e. Arterial thromboembolic events within 6 months prior to first dose, venous thromboembolic events ≥ Grade 3 according to NCI CTCAE v5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy; current hypertension with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg despite oral antihypertensive therapy; f. Receipt of live attenuated vaccines within 28 days; g. Active hepatitis B (defined as HBsAg positive and HBV-DNA ≥ 500 IU/mL); h. Hepatitis C (defined as HCV-RNA positive) i. History of tuberculosis infection or treatment within 1 year prior to signing informed consent; j. Major surgery within 28 days; k. Severe infection within 4 weeks prior to first dose, l. Prior allogeneic bone marrow transplantation or solid organ transplantation; m. Hemoptysis within 2 months prior to signing informed consent with maximum daily volume ≥ 2.5 mL; clinically significant bleeding event; n. Coagulation abnormalities; o. Peripheral neuropathy ≥ Grade 2 according to NCI CTCAE v5.0. p. Concurrent infectious diseases considered unsuitable for participation in the study.

  3. Study Treatment-Related Criteria:

  a. Treatment with systemic immune-stimulatory agents within 4 weeks prior to first dose; b. Treatment with systemic immunosuppressive agents within 2 weeks prior to first dose, c. Known allergy to the investigational drug or any of its excipients; or history of severe allergic reactions to monoclonal antibodies;

  4. Participation in any other clinical trial involving investigational drugs within 4 weeks prior to first dose, or less than five elimination half-lives since last investigational drug administration

  5. History of substance abuse, alcoholism, or illicit drug use

  6. Pregnant, lactating, or planning to become pregnant during the study period

  7. Other serious physical or psychiatric illnesses or laboratory abnormalities that may increase the risk of participation, interfere with the study treatment or results, or in the opinion of the investigator, make the subject unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate (pCR) | Up to approximately 24 weeks
  the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery

SECONDARY OUTCOMES:
Event-free Survival (EFS) as assessed by Investigator | At least 2 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Disease-free Survival (DFS) as assessed by Investigator | At least 2 years
  DFS is defined as the time from surgery to any of the following events: local or distant recurrence, or death due to any cause.
Distant Disease-free Survival (DDFS) as assessed by Investigator | At least 2 years
  DDFS is defined as the time from surgery to distant recurrence, or death due to any cause.
Objective response rate (ORR) in accordance with RECIST v1.1 | Up to approximately 24 weeks
  Number of responders Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed by MRI.
Adverse Events (AEs) | up to 90 days after last dose of ivonescimab
  Incidence rate of AEs of any cause will be evaluated in participants in the Safety Run-In according to CTCAE v5.0.

IPD SHARING:
Plan to Share IPD: Undecided